CLINICAL TRIAL: NCT01079208
Title: Assessment of Growth of Infants Fed Starter Formulas With Modified Protein and Synbiotics
Brief Title: Growth of Infants Fed New Starter Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09.04.INF
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2013-10

CONDITIONS: Dietary Intervention
Keywords: infant formula, synbiotics, probiotics, nutrition
MeSH Terms: interventions — Synbiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- standard starter infant formula (Placebo Comparator): standard starter infant formula
  Interventions: Other: control standard formula
- test starter formula (Experimental): test infant formula
  Interventions: Other: test starter infant formula
- test starter formula with synbiotics (Experimental): starter formula with synbiotics and adapted protein levels
  Interventions: Other: test starter infant formula with synbiotics

INTERVENTIONS:
Other: test starter infant formula — infants are fed for 6 months with this starter formula
  Arms: test starter formula
Other: test starter infant formula with synbiotics — infant are fed for 6 months with this formula
  Arms: test starter formula with synbiotics
Other: control standard formula — infant are fed 6 months with this formula
  Arms: standard starter infant formula

SUMMARY:
The purpose of this study is to assess the growth of infants fed a novel starter formula containing synbiotics and different protein levels, compared to a standard starter infant formula, during the first four months of life.

DETAILED DESCRIPTION:
Breastfeeding represents the "gold standard" for infant health, and efforts are being made to support breast feeding at both the international and local levels. After breast milk, infant formulas are the next best source of nutrition for newborn and growing infants. Science and industry are striving to develop formulas that mimic as close as possible the physiological responses to human milk. There are a multitude of factors that make human milk the physiologically ideal for the infant. Among these, two important factors are the level of protein and the presence of pre-and probiotics in breast milk.

The purpose of this study will be to evaluate growth of healthy infants fed a partially hydrolyzed whey protein formula with a level of protein closer to breast milk, with or without synbiotics, during the first four months of life as compared to the growth of infants fed a partially hydrolyzed whey protein formula with a standard protein level (standard formula). Additionally, the infant's digestive tolerance of the starter formula and frequency of morbidity will be investigated until 6 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborn infant
* Full-term (> 37 weeks gestation)
* Birth weight > 2500 and < 4500 g
* 14±3 days of age on enrollment
* Singleton birth
* Infant's mother has elected not to breastfeed prior to enrollment
* Has not received solid foods
* Having obtained his/her legal representative's informed consent

Exclusion Criteria:

* Known or suspected cow-milk allergy
* Congenital illness or malformation that may affect infant feeding and/or growth
* Significant prenatal and/or postnatal disease
* Any readmission to hospital (except for hyperbilirubinemia) prior to enrollment
* Receiving prescription medication (with exception of treatment for thrush) or frequent use of over the counter medications except vitamin and mineral supplements
* Has received oral or intravenous antibiotic therapy in the last 7 days
* Has received probiotics in the last 7 days
* Currently participating in another clinical study
* Infant's family who in the Investigator's assessment cannot be expected to comply with treatment (feeding regimen)

Ages: 11 Days to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 297 (Estimated)
Dates: Start 2010-03; Primary Completion 2013-12 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Weight gain will be assessed in grams per day, in the period of 14 to 112 days of life (4 months) | 4 months

SECONDARY OUTCOMES:
Tolerance, morbidity, protein status, metabolic markers | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Cabana, MD, MPH, Principal Investigator — Institute for Health Policy Studies, University of California
Locations (3):
- United States (3):
  - UCSF Institute for Health Policy Studies/Pediatrics, San Francisco, California
  - Florida Institute for Clinical Research, Orlando, Florida
  - Midwest Children's Health Research Institute, Lincoln, Nebraska